CLINICAL TRIAL: NCT03576833
Title: The BALLOON- (BALLOon Treatment for Obesity in Norway) Pilot Study
Acronym: BALOON Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Michael Bretthauer, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK 2017/1574
Record Dates: First submitted 2018-06-14; First posted 2018-07-03 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Balloon (Experimental)
  Interventions: Device: Elipse Balloon system

INTERVENTIONS:
Device: Elipse Balloon system — intragastic balloon

SUMMARY:
This protocol describes a feasibility pilot study preceding a randomized clinical study that aims at comparing the Elipse intragastric Balloon system to other invasive obesity techiniques.

The current pilot study is investigating the feasibility and efficacy of the Elipse Balloon system in 20 patients in Norway.

DETAILED DESCRIPTION:
The primary aims of the pilot study are to streamline the infrastructure, machinery, and clinical experience with the balloon before the start of the randomized trial. The inclusion and exclusion criteria, and measurement points will be similar for the two studies.

The primary endpoints of the pilot study are to ascertain the feasibility of

1. Patient recruitment and informed consent process
2. Balloon insertion procedure
3. Follow-up of patients for the period of balloon therapy (one balloon)
4. Data gathering, data management, and endpoint evaluation
5. Adverse event evaluation of balloon insertion and therapy Secondary endpoints are weight loss, HBA1c

Eligible Patients Eligible patients are adults who have been referred for obesity treatment to one of the participating obesity centres and meet all of the inclusion criteria and none of the exclusion criteria.

Inclusion criteria

1. adults 18 year or older with BMI ≥30 and ≤40 kg/m2, and a diagnosis of type 2 diabetes.

Feasibility of the intervention will be assesssed by the investigators. Subjects will be carefully monitored during the study for possible adverse events (AEs) and will be advised to contact the study investigator in case of symptoms of possible adverse events.. During each clinical follow-up visit, the investigator will determine AE occurrences. Each adverse event is considered to be either anticipated or unanticipated as described below.

An AE is any adverse change from the subject's baseline (pre-treatment) condition, including a concurrent illness, occurring during the course of the study whether or not considered related to the study intervention (balloon or surgery). Therefore, an AE can be any unfavorable and/or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the procedure.

All adverse events are described by the local study investigator using the electronic patient record system at the participating site. Adverse events will also be collected once yearly through searches in local and national patient registries (hospital discharge and diagnosis registry, Norwegian cause-of-death registry, Norwegian cancer registry).

AEs are categorized as serious or non-serious. Serious Adverse Event (SAE) are those leading to

* unplanned medical or surgical intervention
* unplanned hospitalization (including emergency department visit)
* prolonged duration of planned hospitalization (>24hrs)
* life threatening illness or injury
* permanent impairment of a body structure or a body function
* Death Planned hospitalization for a pre-existing condition, or a procedure required by the protocol, without serious deterioration in health, is not considered a serious adverse event.

Non-Serious Adverse Events:

Adverse events that do not meet the definition of SAEs.

AE evaluation Each reported SAE is reviewed by an adverse event evaluation committee. The committee consist of three individuals with a medical background relevant for the trial and its interventions. The committee is not blinded to treatment arm as this is not feasible given the nature of the trial interventions and the expected grade of details to review to make a decision. Each member of the AE evaluation committee reviews each case independently. Agreement of whether the SAE is due to the intervention or not (yes, no, An SAE report is submitted to the PIs and the company one time each year during the course of the trial.

Participants will be examined by the study investigators 1 to 3 weeks prior to treatment start (baseline visit), and at weeks 4, 8, 12, 16, 26 and 52 after treatment start.

At the baseline visit, demographic data and medical history is assessed.

All visits include a clinical examination with measurements of body weight, anthropometric measures and blood pressure, laboratory analyses, a registration of supplementation and prescription and over-the-counter drug use, and registration of complications and side effects.

Body weight and composition will be measured with patients wearing light clothing and no shoes using bioelectrical impedance analysis. Anthropometric measures will be recorded with patients in an upright position. Height will be measured using wall mounted stadiometers; waist circumference (WC) will be measured at the point midway between the lowest rib margin and the iliac crest. Height and circumferences will be measured to nearest 0.5 cm and weight to the nearest 0.1 kg.

The following laboratory analysis will be performed: hemoglobin; white blood cell count; platelet count; international normalized ratio; C-reactive protein; blood glucose, HbA1c; insulin, C-peptide; anti-GAD; anti-IA2; sodium; potassium; phosphate; chloride; magnesium; serum iron; ferritin; transferrin; calcium; 1,25 dihydroxyvitamin D; 25 hydroxyvitamin D; parathyroid hormone; thiamine; B12; folate; creatinine; bilirubin; albumin; total protein; alanine aminotransferase; aspartate aminotransferase; alkaline phosphatase A; gamma-glutamyl transpeptidase; amylase; lactate dehydrogenase; triglycerides; total cholesterol; HDL cholesterol; LDL cholesterol; unbound thyroxine; thyroid stimulating hormone;

ELIGIBILITY:
Inclusion Criteria:

* adults 18 year or older with BMI ≥30 and ≤40 kg/m2, and a diagnosis of type 2 diabetes.

Exclusion Criteria:

1. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease
2. Previous bariatric or gastric surgery
3. History of chronic or acute pancreatitis
4. History of small bowel obstructions
5. History of open abdominal and/or pelvic surgery EXCLUDING open appendectomy with a right lower quadrant incision.
6. Thyroid or adrenal disease not controlled with medication
7. History of/or signs and/or symptoms of esophageal, gastric, or duodenal disease such as dysphagia and/or painful swallowing, hiatal hernias >5 centimeter, paraesophageal hernias, chronic or acute inflammation, cancer, varices, diverticula, gastroparesis, ulcers, stricture/stenosis, or achalasia
8. Specific diagnosed genetic or hormonal cause for obesity such as Prader-Willi syndrome
9. Severe coagulopathy, hepatic insufficiency or cirrhosis
10. Unable or unwilling to discontinue use of aspirin and/or non-steroidal anti-inflammatory agents (NSAIDs) at least 14 days prior to Elipse deployment and continuing for 14 days after Elipse excretion
11. Anemia defined as either Hgb <11 g/dL for females and <12 g/dL for males
12. Inability to walk 200 meters without assistance
13. Eating disorders including night eating syndrome (NES), bulimia, or binge eating disorder
14. Current or history of illicit drug use or excessive alcohol use
15. Currently taking the following medications (within 30 days prior to enrolment) and/or anticipated need for these medications during the study: Systemic corticosteroids; anticoagulants (e.g. warfarin, dabigatran) or anti-platelet therapy; narcotics or opiates; anti-seizure medication (e.g. clonazepam, phenytoin)
16. Serum autoantibodies against glutamic acid decarboxylase (GAD) or tyrosine phosphatase (IA2) (MODY or type 1 diabetes)
17. Any specified conditions that, in the opinion of the investigator, may render the subject unable to complete the study without a likely fatal outcome, or lead to difficulties for subject compliance with study requirements, or could confound study data.
18. Women in childbearing age must document a negative pregnancy test. Women must not be breast-feeding at the time of treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Adequate insertion | 4 months
  percentage of adequate balloon insertion and balloon excretion

SECONDARY OUTCOMES:
weight loss | 4 months
  Weight in kg during intervention, and HBA1c values compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided